CLINICAL TRIAL: NCT06548841
Title: Development and Validation of (Bio)Sensors for the Identification of Pathogens
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Tiziana Lazzarotto, Director of the Microbiology Unit - IRCCS Azienda Ospedaliero-Universitaria di Bologna, University of Bologna
Other Study IDs: ECLIPSE
Record Dates: First submitted 2024-07-30; First posted 2024-08-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Infections; Infection, Bacterial; Infection Viral; Infection, Parasite; SARS CoV 2 Infection; Pseudomonas Aeruginosa Infection; Leishmania Infantum Disease
Keywords: infections; platform; nanobiotechnological platforms; bacterial; viral; protozoan; diagnostic; point of care test
MeSH Terms: conditions — Infections; Bacterial Infections; Virus Diseases; Parasitic Diseases; COVID-19; Pseudomonas Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- SARS-CoV2 positive patients: Patients recruited at Personal Genomics (center based in Verona, partner of the European project ECLIPSE), retrospective cohort.
  Interventions: Other: Nanobiotechnology platforms
- SARS-CoV2 negative patients: Patients recruited at Personal Genomics (centre based in Verona), retrospective cohort.
  Interventions: Other: Nanobiotechnology platforms
- P. aeruginosa positive patients: Patients recruited at IRCCS Azienda Ospedaliero-Universitaria di Bologna, prospective cohort.
  Interventions: Other: Nanobiotechnology platforms
- P. aeruginosa negative patients: Patients recruited at IRCCS Azienda Ospedaliero-Universitaria di Bologna, prospective cohort.
  Interventions: Other: Nanobiotechnology platforms
- L. infantum positive patients: Patients recruited at IRCCS Azienda Ospedaliero-Universitaria di Bologna, retrospective and prospective cohort.
  Interventions: Other: Nanobiotechnology platforms
- L. infantum negative patients: Patients recruited at IRCCS Azienda Ospedaliero-Universitaria di Bologna, retrospective and prospective cohort.
  Interventions: Other: Nanobiotechnology platforms

INTERVENTIONS:
Other: Nanobiotechnology platforms — The analyses will be carried out using the novel devices, which are of two types:
  1. The first type of nanobiotechnological platform encompasses the hybridization of pathogen nucleic acids - that may be present in the clinical specimen - by employing specific molecular probes.
  2. The second type of nanobiotechnological platform encompasses the use of capture bacteriophages or "bait Phages" to specifically detect bacterial or protozoan cell surface antigens (in the case of P. aeruginosa or L. infantum respectively) or viral particles (in the case of SARS-CoV2) and the use of reporter bacteriophages ("transducer Phages") for the transduction of the electrochemiluminescent signal.

SUMMARY:
The recent COVID-19 pandemic has revealed the need to develop tests that are accurate, rapid, and inexpensive for the diagnosis of infectious diseases. This problem is relevant not only for viruses, but also for bacteria and parasites: the identification of pathogens at low concentrations by simple and accurate methods is still largely unsatisfied because these microorganisms are structurally complex and are incorporated in composite and diverse biological samples, which can create relevant interferences in pathogens' detection. Direct diagnostic approaches, such as microscopic examination, culture and molecular testing are carried out in equipped laboratories and require long waiting times to obtain the results. Recently developed point-of-care (POC) tests are a group of technologies that miniaturize tests into portable devices such that they can be performed both in well-equipped laboratories and outside the conventional laboratory setting. The present study aims to explore the feasibility and adaptability of newly developed platforms to detect: 1. a virus (SARS-CoV2), 2. a bacterium (Pseudomonas aeruginosa) and 3. a protozoan parasite (Leishmania infantum) in clinical specimens, such as blood and respiratory samples. These newly developed platforms are expected to overcome the current limitations of molecular testing (high cost, time required and need for well-equipped laboratories) and rapid testing (high number of false-negative results). In addition, the newly developed platforms may have important clinical application in low-income countries, which will benefit from a simple and inexpensive approach to detect the many infectious diseases that affect millions of people each year.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining informed consent
* Age ≥ 18 years
* Patients who meet one of the following conditions: SARS-CoV2 positive patients (group 1), SARS-CoV2 negative patients (group 2), P. aeruginosa positive patients (group 3), P. aeruginosa negative patients (group 4), L. infantum positive patients (group 5), L. infantum negative patients (group 6).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: patients with SARS-CoV2 infection. Group 2: patients without SARS-CoV2 infection. Group 3: patients with P. aeruginosa infection. Group 4: patients without P. aeruginosa infection. Group 5: patients with L. infantum infection. Group 6: patients without L. infantum infection.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The evaluation of the sensitivity and specificity of new nanobiotechnological platforms compared to gold standard diagnostic tests | 16 months
  The sensitivity and the specificity will be estimated by creating the confusion matrix corresponding to the classification between signals significant (beyond Limit Of Detection, LOD) and samples giving non-significant signals (below LOD).
  Where the analytical problem is described by other variables than the electrochemiluminescent analytical signal, multivariate classification methods shall be applied. The correlation and interaction between variables will also be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Lazzarotto, PhD, Principal Investigator — University of Bologna, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Department of Medical and Surgical Sciences, University of Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Shared IPD will not include personal data, but will be limited to positive or negative test results to a specific pathogen by employing routine diagnostics techniques and the new devices.
Supporting Information: CSR
Time Frame: Summary data will be published starting 6 months after the end of the study.

REFERENCES:
- [Background] Burrow DT, Heggestad JT, Kinnamon DS, Chilkoti A. Engineering Innovative Interfaces for Point-of-Care Diagnostics. Curr Opin Colloid Interface Sci. 2023 Jun 8:101718. doi: 10.1016/j.cocis.2023.101718. Online ahead of print. PMID 37359425
- [Background] Okeke IN, Ihekweazu C. The importance of molecular diagnostics for infectious diseases in low-resource settings. Nat Rev Microbiol. 2021 Sep;19(9):547-548. doi: 10.1038/s41579-021-00598-5. Epub 2021 Jun 28. PMID 34183821
- [Background] Blann AD, Heitmar R. SARS-CoV-2 and COVID-19: A Narrative Review. Br J Biomed Sci. 2022 Sep 6;79:10426. doi: 10.3389/bjbs.2022.10426. eCollection 2022. PMID 36148046
- [Background] Perveen S, Negi A, Gopalakrishnan V, Panda S, Sharma V, Sharma R. COVID-19 diagnostics: Molecular biology to nanomaterials. Clin Chim Acta. 2023 Jan 1;538:139-156. doi: 10.1016/j.cca.2022.11.017. Epub 2022 Nov 18. PMID 36403665
- [Background] Rossolini GM, Mantengoli E. Treatment and control of severe infections caused by multiresistant Pseudomonas aeruginosa. Clin Microbiol Infect. 2005 Jul;11 Suppl 4:17-32. doi: 10.1111/j.1469-0691.2005.01161.x. PMID 15953020
- [Background] Breidenstein EB, de la Fuente-Nunez C, Hancock RE. Pseudomonas aeruginosa: all roads lead to resistance. Trends Microbiol. 2011 Aug;19(8):419-26. doi: 10.1016/j.tim.2011.04.005. Epub 2011 Jun 12. PMID 21664819
- [Background] Nicoletti G, Schito G, Fadda G, Boros S, Nicolosi D, Marchese A, Spanu T, Pantosti A, Monaco M, Rezza G, Cassone A, Garaci E; CIGAR (Gruppo Cooperativo Infezioni Gravi ed Antibiotico Resistenza). Bacterial isolates from severe infections and their antibiotic susceptibility patterns in Italy: a nationwide study in the hospital setting. J Chemother. 2006 Dec;18(6):589-602. doi: 10.1179/joc.2006.18.6.589. PMID 17267336
- [Background] Buchan BW, Windham S, Balada-Llasat JM, Leber A, Harrington A, Relich R, Murphy C, Dien Bard J, Naccache S, Ronen S, Hopp A, Mahmutoglu D, Faron ML, Ledeboer NA, Carroll A, Stone H, Akerele O, Everhart K, Bonwit A, Kwong C, Buckner R, Warren D, Fowler R, Chandrasekaran S, Huse H, Campeau S, Humphries R, Graue C, Huang A. Practical Comparison of the BioFire FilmArray Pneumonia Panel to Routine Diagnostic Methods and Potential Impact on Antimicrobial Stewardship in Adult Hospitalized Patients with Lower Respiratory Tract Infections. J Clin Microbiol. 2020 Jun 24;58(7):e00135-20. doi: 10.1128/JCM.00135-20. Print 2020 Jun 24. PMID 32350045
- [Background] Burza S, Croft SL, Boelaert M. Leishmaniasis. Lancet. 2018 Sep 15;392(10151):951-970. doi: 10.1016/S0140-6736(18)31204-2. Epub 2018 Aug 17. PMID 30126638
- [Background] Maroli M, Rossi L, Baldelli R, Capelli G, Ferroglio E, Genchi C, Gramiccia M, Mortarino M, Pietrobelli M, Gradoni L. The northward spread of leishmaniasis in Italy: evidence from retrospective and ongoing studies on the canine reservoir and phlebotomine vectors. Trop Med Int Health. 2008 Feb;13(2):256-64. doi: 10.1111/j.1365-3156.2007.01998.x. PMID 18304273
- [Background] Varani S, Cagarelli R, Melchionda F, Attard L, Salvadori C, Finarelli AC, Gentilomi GA, Tigani R, Rangoni R, Todeschini R, Scalone A, Di Muccio T, Gramiccia M, Gradoni L, Viale P, Landini MP. Ongoing outbreak of visceral leishmaniasis in Bologna Province, Italy, November 2012 to May 2013. Euro Surveill. 2013 Jul 18;18(29):20530. PMID 23929116
- [Background] Franceschini E, Puzzolante C, Menozzi M, Rossi L, Bedini A, Orlando G, Gennari W, Meacci M, Rugna G, Carra E, Codeluppi M, Mussini C. Clinical and Microbiological Characteristics of Visceral Leishmaniasis Outbreak in a Northern Italian Nonendemic Area: A Retrospective Observational Study. Biomed Res Int. 2016;2016:6481028. doi: 10.1155/2016/6481028. Epub 2016 Nov 23. PMID 27999807
- [Background] Todeschini R, Musti MA, Pandolfi P, Troncatti M, Baldini M, Resi D, Natalini S, Bergamini F, Galletti G, Santi A, Rossi A, Rugna G, Granozzi B, Attard L, Gaspari V, Liguori G, Ortalli M, Varani S. Re-emergence of human leishmaniasis in northern Italy, 2004 to 2022: a retrospective analysis. Euro Surveill. 2024 Jan;29(4):2300190. doi: 10.2807/1560-7917.ES.2024.29.4.2300190. PMID 38275016
- [Background] Boelaert M, Verdonck K, Menten J, Sunyoto T, van Griensven J, Chappuis F, Rijal S. Rapid tests for the diagnosis of visceral leishmaniasis in patients with suspected disease. Cochrane Database Syst Rev. 2014 Jun 20;2014(6):CD009135. doi: 10.1002/14651858.CD009135.pub2. PMID 24947503
- [Background] Tateo F, Fiorino S, Peruzzo L, Zippi M, De Biase D, Lari F, Melucci D. Effects of environmental parameters and their interactions on the spreading of SARS-CoV-2 in North Italy under different social restrictions. A new approach based on multivariate analysis. Environ Res. 2022 Jul;210:112921. doi: 10.1016/j.envres.2022.112921. Epub 2022 Feb 10. PMID 35150709
- See also: Antimicrobial resistance surveillance in Europe 2023 - 2021 data — http://www.ecdc.europa.eu/en/publications-data/antimicrobial-resistance-surveillance-europe-2023-2021-data
- See also: WHO Regional office for Europe. Manual on case management and surveillance of the leishmaniases in the WHO European Region — http://www.who.int/publications/i/item/9789289052511
- See also: Wehrens R. Chemometrics with R: Multivariate Data Analysis in the Natural Sciences and Life Sciences — http://link.springer.com/10.1007/978-3-642-17841-2

DOCUMENTS (1):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT06548841/Prot_000.pdf